CLINICAL TRIAL: NCT01789749
Title: Soft Coagulation for the Prevention of Adenoma Recurrence After Endoscopic Mucosal Resection (EMR) of Large Sessile Colonic Polyps: A Multicentre, Randomized Trial.
Brief Title: Soft Coagulation for the Prevention of Adenoma Recurrence
Acronym: SCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Michael Bourke (Other)
Responsible Party: Sponsor-Investigator, Professor Michael Bourke, Director of Gastrointestinal Endoscopy, Western Sydney Local Health District
Organization: Western Sydney Local Health District (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HREC/12/WMEAD/139; HREC2012/5/4.6 (3512) (Other: SydneyWAHS HREC - Westmead campus)
Record Dates: First submitted 2012-11-28; First posted 2013-02-12 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Colonic Adenomas
Keywords: snare tip soft coagulation; endoscopic mucosal resection; adenoma recurrence; adenoma; colonoscopy
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients were blinded to the treatment allocation. The endoscopists performing the index and surveillance procedures were not blinded to the treatment.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Coagulation Arm (Active Comparator): Patients do not receive Snare Tip Soft Coagulation to the edge of the endoscopic resection defect
  Interventions: Other: No Snare Tip Soft Coagulation
- Coagulation Arm (Experimental): Patients to receive Snare Tip Soft Coagulation to the edge of the endoscopic resection defect
  Interventions: Other: Snare Tip Soft Coagulation

INTERVENTIONS:
Other: Snare Tip Soft Coagulation
  Arms: Coagulation Arm
Other: No Snare Tip Soft Coagulation
  Arms: No Coagulation Arm

SUMMARY:
Recurrence after endoscopic mucosal resection of laterally spreading lesions (LSL) >= 20mm in size occurs in approximately 20% of cases at surveillance colonoscopy. We aim to evaluate the efficacy of prophylactic adjuvant thermal ablation of the EMR mucosal defect margin in reducing adenoma recurrence following colonic EMR.

ELIGIBILITY:
Inclusion Criteria:

* Referred for removal of a colonic polyp >= 20mm in size
* Able to give informed consent to involvement in trial

Exclusion Criteria:

* Younger than 18 years of age
* Highly dependant on medical care
* Women who are pregnant or may be pregnant.
* Taken clopidogrel within 7 days
* Taken warfarin within 5 days
* Had full therapeutic dose unfractionated heparin within 6 hours
* Had full therapeutic dose low molecular weight heparin (LMWH) within 12 hours
* Known clotting disorder
* Previous attempt at EMR of the polyp referred for resection
* Polyp located at the ileo-caecal valve, appendiceal orifice
* Fully circumferential polyp
* Incomplete snare resection of the polyp

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2013-07; Primary Completion 2016-05-16 (Actual); Study Completion 2016-12-16 (Actual)

PRIMARY OUTCOMES:
Endoscopic recurrence | 4-6 months and 18 months
  Presence of residual/recurrent adenoma at the EMR scar at endoscopic follow-up

SECONDARY OUTCOMES:
Histologic recurrence | 4-6 months and 18 months
  Presence of residual/recurrent adenoma on biopsy of the endoscopic resection scar
En bloc resection | Index procedure
  Rate of 'en bloc resection' (removing entire lesion in one snare) with histologically confirmed clear margins
Snare resections | Index procedure
  The number of snare resections needed to achieve complete clearance
Duration | Index procedure
  Time required for EMR
Perforation during EMR | During index procedure
  Perforation during EMR
Post EMR bleeding | Post Index procedure
  Bleeding after EMR requiring admission or repeat intervention
Number of injections for hemostasis | Index procedure, if post EMR bleeding
  Number of injections required for haemostasis
Location of bleeding vessels | Index procedure, if post EMR bleeding
  Location of bleeding vessels
Size/number of bleeding vessels | Index procedure, if post EMR bleeding
  Size/number of bleeding vessels
Delayed perforation | After index procedure
  Delayed perforation requiring intervention or readmission
Readmission | After index procedure
  Readmission after index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bourke, FRACP, MBBS, Principal Investigator — Western SLHD
Locations (4):
- Australia (4):
  - Westmead Endoscopy Unit, Westmead, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Lyell McEwin Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, VA

REFERENCES:
- [Derived] Klein A, Tate DJ, Jayasekeran V, Hourigan L, Singh R, Brown G, Bahin FF, Burgess N, Williams SJ, Lee E, Sidhu M, Byth K, Bourke MJ. Thermal Ablation of Mucosal Defect Margins Reduces Adenoma Recurrence After Colonic Endoscopic Mucosal Resection. Gastroenterology. 2019 Feb;156(3):604-613.e3. doi: 10.1053/j.gastro.2018.10.003. Epub 2018 Oct 6. PMID 30296436